CLINICAL TRIAL: NCT07318727
Title: Three-Way Diet Comparison for Weight Loss in Overweight Endometrial Cancer Patients on Fertility-Sparing Regimens: A Randomized Controlled Trial
Brief Title: Comparative Study on the Effect of Diet Interventions on Weight Loss in Overweight Endometrial Cancer Patients Undergoing Fertility-sparing Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Li, Director, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHB183-001
Record Dates: First submitted 2024-08-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Endometrium Cancer
Keywords: Endometrial Neoplasms; Dietary Patterns; Body Weight
MeSH Terms: conditions — Endometrial Neoplasms; Body Weight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Fasting Group. (Experimental): Patients in the Intermittent Fasting group used a 5 days in a week are non-fasting days, and the other 2 non-consecutive days are fasting days.
  Interventions: Behavioral: Multi-Professional Guided '5+2' Intermittent Fasting
- Low-energy balanced diet Group. (Experimental): Patients in the Low-energy balanced diet group used the target energy intake for women is 1000-1200 kcal/d. Adopt a balanced diet.
  Interventions: Behavioral: Low-energy Balanced Diet
- Control Group (Other): Patients in the control group underwent routine care for self-weight management.
  Interventions: Behavioral: Routine Care for Self-weight Management.

INTERVENTIONS:
Behavioral: Multi-Professional Guided '5+2' Intermittent Fasting — An intervention team of dietitians, doctors and nurses gave patients specific dietary instructions online and offline. Dietary intervention according to the current research basis, intermittent fasting is mainly adopted, that is, the "5+2 light fasting" mode, in which 5 days in a week are non-fasting days, and the other 2 non-consecutive days are fasting days. The recommended daily energy on non-fasting days is based on body weight: standard body weight (kg) ×20; Or according to body composition measurement lean body mass calculation: BMS =370+21.6× lean body mass (kg), recommended energy intake = BMS × (1.2 ~ 1.3) -500, including protein 20%, fat 25%, carbohydrate 55%. Fasting day energy intake is 1/4 of the usual, about 500 ~ 600kcal.
  Arms: Intermittent Fasting Group.
Behavioral: Low-energy Balanced Diet — The target energy intake for women is 1000-1200 kcal/d. Adopt a balanced diet, in which carbohydrates account for 55% to 60% of the total daily energy, fat accounts for 25% to 30% of the total daily energy, protein 10% to 15%. Increase your intake of fiber-rich, low-energy foods to ensure you feel full.
  Arms: Low-energy balanced diet Group.
Behavioral: Routine Care for Self-weight Management. — The relationship between overweightness and obesity and endometrial cancer risk was explained to patients in the control group and their willingness for self-weight management was respected. Communication was maintained with patients from treatment initiation to 6 and 12 months after treatment; patients' questions regarding weight reduction were answered and suggestions were provided regarding nutrition, exercise, and lifestyle management.
  Arms: Control Group

SUMMARY:
In this study, overweight and obese patients with endometrial cancer treated with fertility- sparing therapy were randomly divided into three groups. The first group was given Intermittent fasting, the second was given Low-energy balanced diet, the third group underwent routine care for self-weight management. Relevant information such as body morphology ,glycolipid metabolism and tumor outcomes of the subjects were collected. By evaluating the tumor outcome and changes in glycolipid metabolism indicators, to confirm the effectiveness and safety of diet interventions for overweight and obese patients with endometrial cancer and treatd with fertility preservation.

DETAILED DESCRIPTION:
Obesity is recognized as a major risk factor for the development of endometrial cancer. Notably, several retrospective studies have shown that obesity reduces complete remission and pregnancy rates and increases recurrence rates in patients with endometrial cancer and atypical hyperplasia who undergo fertility-sparing treatment. Guidelines or consensus statements for fertility sparing treatment in endometrial cancer recommend weight management.The more accepted weight control diet programs mainly include calorie restriction and dietary changes. In dietary management, studies have shown that intermittent fasting ,low-energy balanced diet can improve patient outcomes. This study therefore aimed to investigate the impact of the different dietary interventions on body morphology and composition, glycolipid metabolism, and tumor outcomes in overweight and obese patients with endometrial cancer and atypical hyperplasia who underwent reproductive function-preserving treatments.In this study, overweight and obese patients with endometrial cancer treated with fertility- sparing therapy were randomly divided into second groups. The first group was given Intermittent fasting, the second was given Low-energy balanced diet, the third group underwent routine care for self-weight management.Relevant information such as body morphology ,glycolipid metabolism, molecular typing and tumor outcomes of the subjects were collected. By evaluating the tumor outcome and changes in glycolipid metabolism indicators, to confirm the effectiveness and safety of different dietary interventions management for overweight and obese patients with endometrial cancer and treatd with fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* diagnosed as endometrial cancer or atypical hyperplasia
* fertility-preserving therapy
* BMI≥25 kg/m2
* informed consent.

Exclusion Criteria:

* those with communication barriers
* pregnant women
* medical and surgical serious complications: urinary calculi, history of renal failure or severe renal insufficiency, familial dyslipidemia, severe liver disease, chronic metabolic acidosis, history of pancreatitis, severe diabetes mellitus, active gallbladder disease, fat dyspepsia, severe cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index(BMI) | Baseline /Month 6 of intervention / Month 12 of intervention
  Use the Inbody720 to measure height and weight and calculate BMI according to the formula"BMI (= weight (kg)/height2 (m2)

SECONDARY OUTCOMES:
Complete Pathological Remission of Endometrial Cancer Tumor | Baseline /Month 6 of intervention / Month 12 of intervention
  Defined as the absence of any histological evidence of endometrioid adenocarcinoma or atypical hyperplasia in post-treatment endometrial biopsy or curettage specimens, confirmed by two independent pathologists. This state is characterized by complete regression of the tumor lesion, which may be accompanied by benign findings such as stromal metaplasia or atrophic endometrium
Waist-to-height Ratio(WHtR) | Baseline /Month 6 of intervention / Month 12 of intervention
  Calculate WHtR according to the formula"WHtR= waist circumference (cm)/height (cm)= waist circumference (cm)/height (cm)"
Waist-to-hip Ratio(WHR) | Baseline /Month 6 of intervention / Month 12 of intervention
  Calculate WHR according to the formula"WHR=waist circumference (cm)/hip circumference (cm)"
A Body Shape Index(ABSI) | Baseline /Month 6 of intervention / Month 12 of intervention
  Calculate ABSI according to the formula"ABSI= (waist)/([BMI]^2/3×height^1/2)" Time Frame: 6 months of intervention
Body Roundness Index(BRI) | Baseline /Month 6 of intervention / Month 12 of intervention
  Calculate BRI according to the formula"BRI= waist/BMI" Time Frame: 6 months of intervention
Waist circumference | Baseline /Month 6 of intervention / Month 12 of intervention
  Measured with the subject's body upright, abdomen relaxed, both arms hanging down naturally, feet together, and the tape measure placed around the waist; the height was adjusted to the horizontal plane passing through the midpoint of the line between the lower edge of the rib arch and the iliac crest in the mid-axillary line
Hip circumference | Baseline /Month 6 of intervention / Month 12 of intervention
  Measured with the subject's body upright, taking the circumference of the body at the horizontal position of the uppermost point of the hip
Triglycerides | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Cholesterol | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
High density lipoprotein(HDL) | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Low density lipoprotein | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Fasting glucose | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Fasting insulin | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer
Glycated hemoglobin | Baseline /Month 6 of intervention / Month 12 of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiaodan, Master, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China